CLINICAL TRIAL: NCT00280033
Title: A Randomized, Placebo-Controlled, Phase I/II, Dose-Ranging Study of the Safety, Reactogenicity, and Immunogenicity of Intramuscular Inactivated Influenza A/H5N1 Vaccine Given Alone or Combined With Adjuvants in Healthy Adults
Brief Title: H5 Adult - Chiron Study of Bird Flu Vaccine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 04-062
Record Dates: First submitted 2006-01-19; First posted 2006-01-20 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2009-01

CONDITIONS: Influenza
Keywords: H5N1, Influenza, vaccine, parent protocol
MeSH Terms: conditions — Influenza, Human; Influenza in Birds | interventions — Aluminum Hydroxide; chiron

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (9):
- 9 (Placebo Comparator): Saline administered on days 0 and 28.
  Interventions: Drug: Placebo
- 8 (Experimental): 45 mcg alone administered on days 0 and 28.
  Interventions: Biological: Inactivated Influenza A/H5N1 Vaccine (Chiron)
- 7 (Experimental): 30 mcg plus aluminum hydroxide administered on days 0 and 28.
  Interventions: Biological: Aluminum hydroxide; Biological: Inactivated Influenza A/H5N1 Vaccine (Chiron)
- 6 (Experimental): 30 mcg alone administered on days 0 and 28.
  Interventions: Biological: Inactivated Influenza A/H5N1 Vaccine (Chiron)
- 5 (Experimental): 15 mcg plus aluminum hydroxide administered on days 0 and 28.
  Interventions: Biological: Aluminum hydroxide; Biological: Inactivated Influenza A/H5N1 Vaccine (Chiron)
- 4 (Experimental): 15 mcg plus MF59 administered on days 0 and 28.
  Interventions: Biological: Inactivated Influenza A/H5N1 Vaccine (Chiron); Biological: MF-59
- 3 (Experimental): 15 mcg alone administered on days 0 and 28.
  Interventions: Biological: Inactivated Influenza A/H5N1 Vaccine (Chiron)
- 2 (Experimental): 7.5 mcg plus aluminum hydroxide administered on days 0 and 28.
  Interventions: Biological: Aluminum hydroxide; Biological: Inactivated Influenza A/H5N1 Vaccine (Chiron)
- 1 (Experimental): 7.5 mcg plus MF59 administered on days 0 and 28.
  Interventions: Biological: Inactivated Influenza A/H5N1 Vaccine (Chiron); Biological: MF-59

INTERVENTIONS:
Biological: Aluminum hydroxide — Provided in vials that contain 0.8 mL volume per vial.
  Arms: 2; 5; 7
Biological: Inactivated Influenza A/H5N1 Vaccine (Chiron) — Monovalent subvirion H5N1 vaccine (HA of A/Vietnam/1203/04) provided in unit-dose vials containing 60 mcg/mL A/H5N1 HA as determined by single radial immunodiffusion. It may be formulated with MF59 or aluminum hydroxide. Dosages: 7.5 mcg, 15 mcg, 30 mcg, or 45 mcg.
  Arms: 1; 2; 3; 4; 5; 6; 7; 8
Biological: MF-59 — Proprietary experimental adjuvant. Provided in vials that contain 0.7 mL volume per vial.
  Arms: 1; 4
Drug: Placebo — Saline placebo.
  Arms: 9

SUMMARY:
This study is will gather critical information on the safety, tolerability, and the immunogenicity (capability of causing an immune response) of A/H5N1 (Bird flu) virus vaccine in healthy adults. Up to 400 healthy adults, aged 18 to 64, will participate. Each subject will participate for about 7 months and will be randomly placed in one of several different study groups receiving a different dose of vaccine or placebo. All subjects will receive two injections of their assigned study product, about 28 days apart, in the muscle. Subjects will keep a journal of their temperature and any adverse effects between study visits. A small amount of blood will also be drawn before the first injection, 7 days after each injection, 1 month after the first injection, and 1 and 6 months after the second injection.

DETAILED DESCRIPTION:
The emergence of novel influenza A virus strains in humans (including subtype A/H5N1, H7N7 H9N2 viruses) has added urgency to ongoing efforts to develop plans for responding to potential pandemic situations. This study compares the safety, reactogenicity, and immunogenicity of increasing doses of monovalent subvirion influenza A/H5N1 virus vaccine administered by intramuscular (IM) injection to healthy adults alone or combined with the adjuvants aluminum hydroxide or MF59. The primary objectives are to determine: the dose-related safety of subvirion inactivated H5N1vaccine with and without adjuvants in healthy adults; the dose-related immunogenicity of subvirion inactivated H5N1vaccine with and without adjuvants in healthy adults approximately 1 month following receipt of 2 vaccine doses; to provide information for the selection of the best dosage level for further studies. The secondary objectives are to evaluate dose-related immunogenicity and the percent of subjects responding about 1 and 7 months after the first vaccination. The primary endpoints are: adverse event (AE) or serious adverse event (SAE) information; proportion of subjects in each dose group achieving a serum neutralizing antibody titer of 1:40 against the influenza A/H5N1 virus 28 days after receipt of the second dose of vaccine; proportion of subjects in each dose group achieving a serum hemagglutination (HAI) antibody titer of 1:40 against the influenza A/H5N1 virus 28 days after receipt of the second dose of vaccine; geometric mean titer (GMT) and frequency of 4-fold or greater increases in neutralizing antibody titers in each group 28 days after receipt of the second dose of vaccine; geometric mean titer and frequency of 4-fold or greater increases in serum HAI antibody titers in each group 28 days after receipt of the second dose of vaccine. The secondary endpoints are: GMT and frequency of 4-fold or greater increases in neutralizing antibody titers in each group 1 month and 7 months after receipt of the first dose of vaccine; geometric mean titer and frequency of 4-fold or greater increases in serum HAI antibody titers in each group 1 month and 7 months after receipt of the first dose of vaccine; development of serum antibody responses against antigenically drifted variants of H5N1 influenza virus. The primary outcome measures will be the frequencies and severities of AEs in each group and the proportions of subjects who achieve a serum neutralizing antibody titer of 1:40 against the influenza A/H5N1 virus on Day 56. About 390 healthy adults, 18 to 64 years old, inclusive, will be enrolled into this multicenter, randomized, placebo-controlled, dose-ranging clinical trial. Nine groups of randomized subjects will receive two doses of saline placebo or influenza A/H5N1 vaccine at 45, 30, or 15 micrograms; or influenza A/H5N1 vaccine at 15 or 7.5 micrograms with MF59; or influenza A/H5N1 vaccine with aluminum hydroxide at 30, 15, or 7.5 micrograms (N=30, 60 or 90/vaccine dose group total 390). Laboratory safety profile blood will be drawn prior to the first immunization. Subjects will receive 2 doses approximately 28 days apart. Subjects will be observed after inoculation and maintain a memory aid for 7 days afterwards. Subjects will be telephoned 1 to 3 days after vaccination for AE assessment, and they will return to the clinic on Day 7 for AE and concomitant medication assessment, targeted physical examination, safety laboratory tests and a review of the memory aid. Telephone calls assessing AEs will be performed after each vaccination. Serum for safety laboratory tests will be obtained prior to and approximately 7 days after first and second immunizations. I

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or nonpregnant female (as indicated by a negative urine pregnancy test immediately prior to vaccine administration) between the ages of 18 and 64 years, inclusive.
* Women of childbearing potential (not surgically sterile or post menopausal for greater than or equal to one year) must agree to practice adequate contraception (i.e., barrier method, abstinence, and licensed hormonal methods) for the entire study period.
* Is in good health, as determined by vital signs (heart rate, blood pressure, oral temperature), medical history and a targeted physical examination based on medical history.
* Subjects should have normal safety laboratory values (Hgb, WBC, Plt, ALT, and creatinine) prior to the first immunization.
* Able to understand and comply with planned study procedures.
* Provides written informed consent prior to initiation of any study procedures.

Exclusion Criteria:

* Has a known allergy to eggs or other components of the vaccine or latex.
* Has a positive urine pregnancy test prior to vaccination (if female of childbearing potential) or women who are breastfeeding.
* Is undergoing immunosuppression as a result of an underlying illness or treatment.
* Has an active neoplastic disease or a history of any hematologic malignancy.
* Is using oral or parenteral steroids, high-dose inhaled steroids (greater than 800 micrograms/day of beclomethasone dipropionate or equivalent) or other immunosuppressive or cytotoxic drugs (nasal and topical steroids are allowed).
* Has a history of receiving immunoglobulin or other blood products within the 3 months prior to vaccination in this study.
* Has received any other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to vaccination in this study.
* Has an acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the evaluation of responses (this includes, but is not limited to: known chronic liver disease, significant renal disease, unstable or progressive neurological disorders, diabetes mellitus, and transplant recipients).
* Has a history of severe reactions following immunization with contemporary influenza virus vaccines.
* Has an acute illness, including an oral temperature greater than 100.4 degrees F, within 1 week of vaccination.
* Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to vaccination in this study, or expects to receive an experimental agent during the 7-month study period.
* Has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.
* Participated in H5 vaccine study in the past.
* Known current HIV, hepatitis B (HBsAg) or hepatitis C infection.
* History of alcohol or drug abuse in the last 5 years.
* Planned travel outside the US between vaccination and the second study visit.
* History of Guillain-Barre.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 394 (Actual)
Dates: Start 2006-02; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Geometric mean titer and frequency of 4-fold or greater increases in serum hemagglutination inhibition (HAI) antibody titers in each group 28 days after receipt of the second dose of vaccine. | Approximately Day 56.
Adverse event or SAE information (solicited in-clinic and via memory aids, concomitant medications, and periodic targeted physical assessments). | Adverse events will be collected through 28 days following the second dose of vaccine (approximately Day 56). Serious adverse events will be collected throughout the study through Day 208.
Proportion of subjects in each group achieving a serum neutralizing antibody titer ratio of 1:40 against the influenza A/H5N1 virus 28 days following second dose of vaccine. | Approximately Day 56.
Proportion of subjects in each dose group achieving a serum hemagglutination (HAI) antibody titer of 1:40 against the influenza A/H5N1 virus 28 days after receipt of the second dose of vaccine. | Approximately Day 56.
Geometric mean titer (GMT) and frequency of 4-fold or greater increases in neutralizing antibody titers in each group 28 days after receipt of the second dose of vaccine. | Approximately Day 56.

SECONDARY OUTCOMES:
Geometric mean titer and the frequency of 4-fold or greater increases in neutralizing antibody titers in each group 1 month after receipt of each dose, and 7 months after receipt of the first dose of vaccine. | Blood samples for serum assays will be collected at Day 0 and at Days 28, 56, and 208 after the first immunization.
Geometric mean titer and the frequency of 4-fold or greater increases in serum HAI antibody titers 1 month after receipt of each dose, and 7 months after receipt of the first dose of vaccine. | Blood samples for serum assays will be collected at Day 0 and at Days 28, 56, and 208 after the first immunization.
Development of serum antibody responses against antigenically drifted variants of H5N1influenza virus. | Blood samples for serum assays will be collected at Day 0 and at Days 28, 56, and 208 after the first immunization.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Stanford University, Stanford, California
  - Saint Louis University, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Vanderbilt University, Nashville, Tennessee

REFERENCES:
- [Result] Bernstein DI, Edwards KM, Dekker CL, Belshe R, Talbot HK, Graham IL, Noah DL, He F, Hill H. Effects of adjuvants on the safety and immunogenicity of an avian influenza H5N1 vaccine in adults. J Infect Dis. 2008 Mar 1;197(5):667-75. doi: 10.1086/527489. PMID 18260764